CLINICAL TRIAL: NCT01390454
Title: Study of the Relationship Between Functional Ultrasound Data and the Impact of Lateral Epicondylar Pain
Brief Title: Relationships Between Ultrasound Data and the Impact of Lateral Epicondylar Pain
Acronym: EPICORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2010/AD-03b; 2011-A00769-32 (Other: RBC number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Tennis Elbow; Epicondylitis, Lateral Humeral
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tennis elbow patients (Experimental): These patients have tennis elbow, according to stated inclusion criteria.
  Interventions: Procedure: Ultrasound of the elbow 1, days 7 to 15; Procedure: Ultrasound of the elbow 2, days 7 to 15; Procedure: Ultrasound of the elbow 3, days 45 to 90
- Healthy volunteers (Active Comparator): Healthy volunteers are selected and paired according to age, sex, socio-professional category and left- or right-handedness.
  Interventions: Procedure: Ultrasound of the elbow 1, days 7 to 15; Procedure: Ultrasound of the elbow 2, days 7 to 15

INTERVENTIONS:
Procedure: Ultrasound of the elbow 1, days 7 to 15 — The primary endpoint is evaluated a first time via an ultrasound exam.
Procedure: Ultrasound of the elbow 2, days 7 to 15 — The primary endpoint is evaluated a second time by a second practitioner.
Procedure: Ultrasound of the elbow 3, days 45 to 90 — A third ultrasound is performed only on tennis elbow patients between days 45 and 90.
  Arms: Tennis elbow patients

SUMMARY:
Our primary objective is to study the relationship between ultra sound data and the pain associated with tennis elbow.

ELIGIBILITY:
Inclusion Criteria for Tennis Elbow patients:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 90 days of follow up
* Pain when pressure applied to the epicondyl
* Pain upon forced movement of both epicondylien muscles
* Absence of pain upon forced movement of an epitrochlear muscle
* Absence of one or more skeletal-muscle problem on the homolateral arm felt by the patient to be just as problematic as his/her tennis elbow
* at least one consult for pain treatment associated with tennis elbow (on the same elbow)

Inclusion Criteria for healthy volunteers:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* No pain when pressure applied to the epicondyl
* No pain upon forced movement of both epicondylien muscles
* No neck pain
* No skeletal-muscle problems in the arms during the 3 months preceding the study

Exclusion Criteria for Tennis Elbow patients:

* The patient is included in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* Absence of one or more skeletal-muscle problem on the homolateral arm felt by the patient to be just as problematic as his/her tennis elbow

Exclusion Criteria for Health Volunteers:

* The subject is included in another study
* The subject is in an exclusion period determined by a previous study
* The subject is under judicial protection, under tutorship or curatorship
* The subject refuses to sign the consent
* It is impossible to correctly inform the subject
* Presence of one or more skeletal-muscle problems in the arms within the 3 months preceding the study
* Pain when pressure applied to the epicondyl
* Pain upon forced movement of both epicondylien muscles
* Consultation for any kind of treatment for elbow pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2013-06-18 (Actual); Study Completion 2013-06-18 (Actual)

PRIMARY OUTCOMES:
Epicondylar surface movement relative to the supinators - extensor carpi radialis brevis and longus (affected elbow) | Days 7 to 15
  The movement of the superficial epicondyliens relative to the supinator is studied via ultrasound and classified as follows: A) good interface movement in both directions; B) good movement in only 1 direction; C) bad movement over less than half of the interface; D) bad movement over a majority of the interface; E) no movement along the interface.
Epicondylar surface movement relative to the supinators - extensor carpi radialis brevis and longus (good elbow) | Days 7 to 15
  The movement of the superficial epicondyliens relative to the supinator is studied via ultrasound and classified as follows: A) good interface movement in both directions; B) good movement in only 1 direction; C) bad movement over less than half of the interface; D) bad movement over a majority of the interface; E) no movement along the interface.

SECONDARY OUTCOMES:
Visual Analog Scale for pain | Baseline
  A visual analog scale ranging from 0 to 100 is used to evaluate pain.
Visual Analog Scale for pain | Between days 45 and 90
  A visual analog scale ranging from 0 to 100 is used to evaluate pain.
Q-Dash Questionnaire | Baseline
  The Quick DASH questionnaire is used to evaluate functional changes.
Q-Dash Questionnaire | Between 45 and 90 days
  The Quick DASH questionnaire is used to evaluate functional changes.
Thickness of the ECR longus and ECR brevis interface | Between days 7 and 15
  The thickness of the interface between the extensor carpi radialis (ECR) longus and the extensor carpi radialis brevis is measured during the ultrasound (mm)
Thickness of the ECR longus and ECR brevis interface, tennis elbow patients only | Between days 45 and 90
  The thickness of the interface between the extensor carpi radialis (ECR) longus and the extensor carpi radialis brevis is measured during the ultrasound (mm)
Thickness of the ECR -supinator interface | Between 7 and 15 days
  The thickness of the intersection (at the base) between the Extensor Carpi Radialis (ECR) muscles and the supinator is measured during ultrasound (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, France